CLINICAL TRIAL: NCT04372784
Title: A Randomized Controlled Trial of Cryotherapy on Benign Anastomotic Strictures Following Esophagectomy, Gastrectomy, and Bariatric Surgery
Brief Title: Cryoablation for Benign Gastrointestinal Anastomotic Strictures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Kulmeet Sandhu, Clinical Associate Professor of Surgery, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HS-19-00679
Record Dates: First submitted 2020-04-29; First posted 2020-05-04 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Esophageal Stricture; Duodenal Stricture; Jejunal Stricture; Anastomotic Stricture of Small Intestine
MeSH Terms: conditions — Esophageal Stenosis | interventions — Cryotherapy; Endoscopy, Digestive System

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- EGD with Balloon Dilatation (Active Comparator): Esophagogastroduodenoscopy with balloon dilatation
  Interventions: Procedure: Esophagogastroduodenoscopy with Balloon Dilatation
- EGD with Balloon Dilatation and Cryotherapy (Experimental): Esophagogastroduodenoscopy with balloon dilatation and cryotherapy
  Interventions: Device: Cryotherapy; Procedure: Esophagogastroduodenoscopy with Balloon Dilatation

INTERVENTIONS:
Device: Cryotherapy — Cryotherapy entails introducing a 9 French catheter via the endoscope's accessory port. The catheter is advanced until it is visualized on the endoscopy monitor. Under 4 psi pressure, liquid nitrogen is sprayed from the catheter for twenty seconds over each four-centimeter segment of stricture
  Arms: EGD with Balloon Dilatation and Cryotherapy
Procedure: Esophagogastroduodenoscopy with Balloon Dilatation — This procedure entails deploying a balloon via the accessory port of the esophagogastroduodenoscope under direct visualization and serially inflating the balloon. Balloon dilatation disrupts not only the muscular rings surrounding strictures but also the granulation tissue composing the strictures.

SUMMARY:
Anastomotic stricture is a common complication following foregut surgery. The standard of care for these benign foregut anastomotic strictures is balloon dilatation. However, re-stenosis of strictures is also common, requiring frequent repetition of balloon dilatation. Cryotherapy is a novel therapy that may improve clinical outcomes following dilatation. The purpose of the present study is to conduct a randomized controlled trial to characterize the impact of cryotherapy on clinical outcomes and complications for benign anastomotic strictures following esophagectomy, gastrectomy, and bariatric surgery.

ELIGIBILITY:
Inclusion Critieria

* History of esophagectomywith primary anastomosis
* History of gastrectomy with primary anastomosis
* History of bariatric surgery with primary anastomosis
* History of anastomotic stricture
* History of balloon dilatation at Keck Hospital of the University of Southern California

Exclusion Critieria

* Patients treated at medical centers other than Keck Hospital of the University of Southern California
* History of anastomotic stent placement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Number of Dilatations | One year
  Total number of dilations within one year

SECONDARY OUTCOMES:
Dilatation size | Immediately after the intervention/procedure/surgery/etc
  Dilatation size (as a proportion to size at presentation)
Perforation rate | Immediately after the intervention/procedure/surgery/etc
  Rates of hollow viscus perforation
Bleeding rate | Immediately after the intervention/procedure/surgery/etc
  Rates of clinically significant bleeding
Fistula rate | One year
  Rates of fistula formation
Reintervention | One year
  Rates of unplanned reintervention (e.g., stenting)
Readmission | One year
  Rates of readmission

CONTACTS AND LOCATIONS:
Locations (1):
- Keck Hospital of USC, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting six months after study publication